CLINICAL TRIAL: NCT04325997
Title: Applicaion of Mouth Opener Combined With Electronic Video Laryngoscope in Double-lumen Intubation of Patients With Difficult Airway
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zhuan Zhang (Other)
Responsible Party: Sponsor-Investigator, Zhuan Zhang, Clinical Professor, Yangzhou University
Organization: Yangzhou University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 20200207
Record Dates: First submitted 2020-02-08; First posted 2020-03-30 (Actual); Last update posted 2020-03-30 (Actual); Status verified 2020-02

CONDITIONS: Difficult Airway Intubation; Double-lumen Tube
Keywords: video laryngoscop; double-lumen tube; mouth gag
MeSH Terms: interventions — Laryngoscopes

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- an ordinary laryngos with mouth opener (Experimental)
  Interventions: Device: laryngoscope with mouth opener
- Video laryngoscopy intubation (No Intervention)
- Video laryngoscope with mouth opener (Experimental)
  Interventions: Device: video laryngoscope with mouth opener

INTERVENTIONS:
Device: laryngoscope with mouth opener — Double-lumen tube combined with mouth gag for laryngoscope intubation
  Arms: an ordinary laryngos with mouth opener
Device: video laryngoscope with mouth opener — Double-lumen tube combined with mouth gag for video laryngoscope intubation
  Arms: Video laryngoscope with mouth opener

SUMMARY:
How to quickly expose glottis and accurately insert double luminal tracheal tube in patients with difficult airway in thoracoscopic surgery has become an urgent problem in anesthesia induction.This study through the double cavity bronchial tube visual laryngoscope intubation with open mouth and electronic video laryngoscope used in combination, to explore whether can shorten the glottis exposure, improve the success rate of the double lumen tube intubation will reduce pharyngeal damage, reduce intubation hemodynamic fluctuations, in order to improve the glottis appeared difficult patients with bronchial intubation success rate to provide the reference.

DETAILED DESCRIPTION:
A total of 60 patients who needed double-lumen endobronchial catheterization in thoracic department and whose Arne o 'risk index score was at least 7 points were randomly divided into three groups.Group B was intubated with video laryngoscopy.Group C was intubated with a mouth opener for video laryngoscope combined with a double-lumen bronchial tube for video laryngoscope intubation (hereinafter referred to as the mouth opener).The glottis exposure time, bronchial intubation time, intubation times, success rate of one intubation, and NRS score of pharyngeal pain 8 hours after surgery were observed and recorded in the three groups, and the hemodynamic changes after intubation were observed and recorded.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of early lung cancer
* Ages ranged from 30 to 80

Exclusion Criteria:

* Pregnancy
* Prediction of difficulty in mask ventilation
* Chest X-ray examination of trachea, bronchial anatomical abnormalities or tumor compression caused by trachea/bronchial deformation
* Failure of assessing Arne risk index

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2019-08-30 (Actual); Study Completion 2019-08-30 (Actual)

PRIMARY OUTCOMES:
Glottis exposure time | through study completion, an average of 1 minute
Bronchial intubation time | through study completion,an average of 1 minute
The number of intubation | through study completion,an average of 1 minute
One-time success rate of intubation | through study completion,an average of 1 minute
Glottic field grading | through study completion,an average of 1 minute
  Cormack-Lehane grading, C-L1：Can see glottis mostly；C-L2：Only the posterior union of the glottis is visible, not the glottis, and at most the cartilago arytaenoidea is visible when the larynx is lightly pressed；C-L3： can't see any part of the glottis, only the epiglottis； C-L4：No part of the larynx can be seen

CONTACTS AND LOCATIONS:
Locations (1):
- the Affiliated Hospital of Yangzhou University, Yangzhou, Jiangsu, China